CLINICAL TRIAL: NCT02386358
Title: Etiologic Treatment With Benznidazole in Adult Patients With Chronic Chagas Disease. A Randomized Double Blind Clinical Trial
Brief Title: Etiologic Treatment With Benznidazole in Adult Patients With Chronic Chagas Disease. A Randomized Clinical Trial
Acronym: TRAENA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Parasitologia Dr. Mario Fatala Chaben (Other Government)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government); Pan American Health Organization (Other); Becas Carrillo Oñativia, Ministerio de Salud, Argentina (Unknown); Drugs for Neglected Diseases (Other)
Responsible Party: Principal Investigator, Adelina Rosa Riarte, Adelina Rosa Riarte MD, Instituto Nacional de Parasitologia Dr. Mario Fatala Chaben
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRAENA
Record Dates: First submitted 2015-01-19; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Chagas Disease
Keywords: Chronic Chagas Disease; Randomized Clinical Trial double blind; Benznidazole vs Placebo; Adult patients
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Benznidazole (Active Comparator): Benznidazole pills of 100 mg, dose 5 mg/Kg/day, twice a day during 60 days
  Interventions: Drug: Benznidazole
- Placebo (Placebo Comparator): Placebo pills 100 mg, dose 5mg/Kg/day, twice a day, during 60 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benznidazole — Benznidazole at a dose 5 mg/Kg/day until 60 days have been completed or development of non-acceptable toxicity-
  Other Names: Radanil (Roche Laboratory)
  Arms: Benznidazole
Drug: Placebo — Placebo at a dose 5 m/Kg/day until 60 days
  Other Names: Placebo pills
  Arms: Placebo

SUMMARY:
The purpose of this study is:

1. -to determine whether benznidazole (BZN) will be able to modify the natural evolution of chronic Chagas disease in adult patients by means of a randomized, double-blind clinical trial (RCT).

   Also:
2. -to validate therapeutic efficacy with new methods, such as recombinant antigen F29 of Trypanosoma cruzi visualized by conventional ELISA, in the context of the RCT compared with conventional serology (CS)
3. -to develop the real-time polymerase chain-reaction (RT-PCR) to quantify the parasite load as an early therapeutic effect.
4. to determine the potential of such serological and parasitological methods as predictors of therapeutic effect or failure.

DETAILED DESCRIPTION:
Patients and Methods. Patients selected to be enrolled were born in Chagas disease endemic areas of Argentina and bordering countries such as Bolivia and Paraguay, whose current residence is in urban non endemic areas of Argentina. They were sorted by clinical stage: stage 0, 1, 2 and 3 according to a modified Kuschnir classification.1 Briefly, Stage 0 corresponds to patients only with reactive serology for Chagas disease; stage 1, patients with reactive serology plus electrocardiographic abnormalities; stage 2, patients with the abovementioned characteristics plus dilatation of left ventricle by echocardiography, and stage 3, patients with the abovementioned characteristics, plus cardiac failure.

The follow-up was performed every 4 months during the first 2 years, every 6 months in the 3rd and 4th year, and annually from then on until the end of the study in 2012.

The safety of TRAENA was controlled at days 25 and 45 intra-treatment by means of laboratory tests and clinical evaluation, and at any time that an adverse event was apparent in patients.

Adherence to medication administration was verified by means of a booklet where the patient recorded the daily intake of medication and any physical abnormality that appeared during the time they were taking of medicine. Adherence was controlled by a surveillance and recovery system which consisted of telephone calls, telegrams, letters or home visits that was termed "active monitoring", which was immediately applied to the control visit when the patient did not attend the corresponding schedule control.

Telephone calls were the most useful tool to recover adherence to monitoring. Patients were assigned to BZN or Placebo treatment by an investigator independent from the research group. Prior to randomization, a pre randomization stratification was performed according to prognostic factors based on clinical stages of Chagas disease.

A database was designed to be used as the registry for the whole study. Demographic, epidemiologic, serologic, parasitological and clinical variables were used in its design, and were registered pre treatment, intra treatment and post treatment throughout the monitoring. Medical records were the primary documents for the registry, where all the variables were recorded manually. Based on the data, variables were registered on a daily basis and a random weekly check was conducted on the data against the medical records. Our Standard Operating Procedure was based on the following procedures: patient screening, selection and coding, sample collection, serum bank, DNA sample storage, monitoring systematization, surveillance systems to recover patients who had discontinued monitoring, etc.

In October 2011 the Base Data Monitoring Board for the last Interim Analysis, recommended an addendum modifying the secondary outcomes, adding simple and combined events. These events were characterized only by electrocardiographic abnormalities or associated to echocardiographic ones. These events were evaluated up April 2013.

ELIGIBILITY:
Inclusion Criteria:

* Patients living in urban areas
* Reactive to at least 2 for serological test performed in Fatala Chaben Institute (ELISA and IFI) ,
* Patients who agreed to be part of this protocol through informed consent form signed

Exclusion Criteria:

* Patients with chronic Chagas disease who have received prior treatment with benznidazole
* Other cardiomyopathies : idiopathic , alcoholic , peripartum myocarditis, secondary to coronary artery disease, valve disease, hypertension, restrictive, hypertrophic or congenital
* Chronic renal disease
* Bleeding disorders
* History of liver disease or current liver disease ,
* Any other severe clinical disease that decreases their life expectancy
* History of severe allergies
* Pregnant patients
* Patients who have not signed the informed consent.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 910 (Actual)
Dates: Start 1999-03; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Mortality | Time to event: from date of randomization until the date of first documented progression or date of death from any cause up to 10 years of follow-up
  Sudden death, unexpectedly in time and in its presentation,preceded by the abrupt loss of consciousness within a maximum of one hour of the onset of symptoms,when it happened during sleep or unexpectedly in a patient was stable until then. Related Death, when presented in a patient with signs of progressive heart failure.Ischemic or Hemorrhagic Stroke
Development of heart failure | Time to event: from date of randomization until the date of first documented progression of heart failure up to 10 years of follow-up
  Dyspnea is evaluated according to the classification of the New York Heart Association (NYHA),gallop rhythm, jugular venous distension, crackles in the lungs, edema or pleural effusion,hepatomegaly
Severe arrhythmias with hemodynamic compromise or pacemaker implant or Implantable cardiac defibrillator | Time to event: from date of randomization until the date of first documented progression up to 10 years of follow-up
  Sustained ventricular tachycardia, atrioventricular block, trifascicular block, Atrial fibrillation

SECONDARY OUTCOMES:
Electrocardiographic endpoints. New development of permanent changes in the electrocardiographic | Time to event: from date of randomization until the date of first documented as defined in the secondary outcome up to 10 years of follow-up
  * Stable sinus bradycardia (<50 beats / min)
  * Auriculoventricular blocks of 2nd and 3rd degree
  * Left anterior hemi-block
  * Complete right bundle branch block
  * Atrial flutter or fibrillation
  * Sustained ventricular tachycardia
Changes in clinical stage in chronic Chagas disease | Time to event: from date of randomization until the date of first documented as defined in the secondary outcome up to 10 years of follow-up
  Clinical progression
Enlargement of the left ventricle (LV) detected by echocardiography. | Time to event: from date of randomization until the date of first documented as defined in the secondary outcome up to 10 years of follow-up
  Clinical Progression
New Heart Failure | Time to event: from date of randomization until the date of first documented as defined in the secondary outcome up to 10 years of follow-up
  Clinical Progression
Stroke | Time to event: from date of randomization until the date of first documented as defined in the secondary outcome up to 10 years of follow-up
  Clinical progression
Serological negativization | time to event: from the date of randomization to the date of the first documented serological negativization that persists until 10 years of follow-up
  by ELISA F29 vs. conventional serology as a late indicator of efficacy or therapeutic failure.
Development and validation of RT-PCR | time to event: from the date of randomization to the date of the first documented no detectable RT-PCR that persists until 10 years of follow-up
  Demonstration of RT-PCR as an early indicator of efficacy or therapeutic failure.
Changes of the secondary objectives during RCT development. New single endpoints | Since October 2011 during 18 months
  1. Any change in clinical stage 0 to II due to left ventricular enlargement demonstrated by echocardiogram, or I to III stage due to development of heart failure.
  2. Complete left branch block
     * 3. Atrial fibrillation
     * 4. Repetitive ventricular extrasystoles: doublets, triplets, bigemina, trigeminus, ventricular tachycardia
Combined clinical endpoints: | Since October 2011 during 18 months
  * Right bundle branch block associated with left anterior hemi-block.
  * Parietal motility disorders of left ventricle by echocardiography (akinesia, hypokinesia, and dyskinesia) associated with impaired left ventricular systolic function.
  * Parietal motility disorders of left ventricle by echocardiogram (Akinesia, Hypokinesia, dyskinesia) and /or impaired LV systolic function associated with new electrocardiographic changes (complete left branch block, right bundle branch block, left anterior hemi-block, ventricular extrasystoles.
  * Occurrence of left ventricle aneurysm point by echocardiogram associated to ventricular arrhythmia (section 2.4.1.4.).
  * Occurrence of left ventricle aneurysm point by echocardiogram associated with depression of LV systolic function by echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Adellina R Riarte, MD, Principal Investigator — Chief of Clinical, Pathology and Treatment Department
Locations (1):
- Instituto Nacional de Parasitología Dr Mario Fatala Chaben, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Result] Sosa Estani S, Segura EL, Ruiz AM, Velazquez E, Porcel BM, Yampotis C. Efficacy of chemotherapy with benznidazole in children in the indeterminate phase of Chagas' disease. Am J Trop Med Hyg. 1998 Oct;59(4):526-9. doi: 10.4269/ajtmh.1998.59.526. PMID 9790423
- [Result] de Andrade AL, Zicker F, de Oliveira RM, Almeida Silva S, Luquetti A, Travassos LR, Almeida IC, de Andrade SS, de Andrade JG, Martelli CM. Randomised trial of efficacy of benznidazole in treatment of early Trypanosoma cruzi infection. Lancet. 1996 Nov 23;348(9039):1407-13. doi: 10.1016/s0140-6736(96)04128-1. PMID 8937280
- [Result] Viotti R, Vigliano C, Armenti H, Segura E. Treatment of chronic Chagas' disease with benznidazole: clinical and serologic evolution of patients with long-term follow-up. Am Heart J. 1994 Jan;127(1):151-62. doi: 10.1016/0002-8703(94)90521-5. PMID 8273735
- [Result] Viotti R, Vigliano C, Lococo B, Bertocchi G, Petti M, Alvarez MG, Postan M, Armenti A. Long-term cardiac outcomes of treating chronic Chagas disease with benznidazole versus no treatment: a nonrandomized trial. Ann Intern Med. 2006 May 16;144(10):724-34. doi: 10.7326/0003-4819-144-10-200605160-00006. PMID 16702588
- [Result] Porcel BM, Bontempi EJ, Henriksson J, Rydaker M, Aslund L, Segura EL, Pettersson U, Ruiz AM. Trypanosoma rangeli and Trypanosoma cruzi: molecular characterization of genes encoding putative calcium-binding proteins, highly conserved in trypanosomatids. Exp Parasitol. 1996 Dec;84(3):387-99. doi: 10.1006/expr.1996.0127. PMID 8948328
- [Result] Kuschnir E, Sgammini H, Castro R, Evequoz C, Ledesma R, Brunetto J. [Evaluation of cardiac function by radioisotopic angiography, in patients with chronic Chagas cardiopathy]. Arq Bras Cardiol. 1985 Oct;45(4):249-56. No abstract available. Spanish. PMID 3835868
- [Result] Reyes PA, Vallejo M. Trypanocidal drugs for late stage, symptomatic Chagas disease (Trypanosoma cruzi infection). Cochrane Database Syst Rev. 2005 Oct 19;(4):CD004102. doi: 10.1002/14651858.CD004102.pub2. PMID 16235350
- [Result] Villar JC, Perez JG, Cortes OL, Riarte A, Pepper M, Marin-Neto JA, Guyatt GH. Trypanocidal drugs for chronic asymptomatic Trypanosoma cruzi infection. Cochrane Database Syst Rev. 2014 May 27;2014(5):CD003463. doi: 10.1002/14651858.CD003463.pub2. PMID 24867876
- [Result] Schijman AG, Bisio M, Orellana L, Sued M, Duffy T, Mejia Jaramillo AM, Cura C, Auter F, Veron V, Qvarnstrom Y, Deborggraeve S, Hijar G, Zulantay I, Lucero RH, Velazquez E, Tellez T, Sanchez Leon Z, Galvao L, Nolder D, Monje Rumi M, Levi JE, Ramirez JD, Zorrilla P, Flores M, Jercic MI, Crisante G, Anez N, De Castro AM, Gonzalez CI, Acosta Viana K, Yachelini P, Torrico F, Robello C, Diosque P, Triana Chavez O, Aznar C, Russomando G, Buscher P, Assal A, Guhl F, Sosa Estani S, DaSilva A, Britto C, Luquetti A, Ladzins J. International study to evaluate PCR methods for detection of Trypanosoma cruzi DNA in blood samples from Chagas disease patients. PLoS Negl Trop Dis. 2011 Jan 11;5(1):e931. doi: 10.1371/journal.pntd.0000931. PMID 21264349
- See also: National Administration of Health Laboratories and Institutes "Dr Carlos G. Malbrán"/ National Institute of Parasitology — http://www.anlis.gov.ar/inp